CLINICAL TRIAL: NCT05061602
Title: Biomechanical and Viscoelastic Properties of Plantar Fascia in Diabetes Mellitus
Acronym: DMumecPRO
Status: Completed | Type: Observational
Sponsor: Tülay Çevik Saldıran (Other)
Collaborators: Okan University (Other)
Responsible Party: Sponsor-Investigator, Tülay Çevik Saldıran, Sponsor-Investigator, Bitlis Eren University
Organization: Bitlis Eren University (Other)
Other Study IDs: BitlisErenUn
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
Keywords: Plantar Fascia; Stiffness; Diabetes mellitus; Fear
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Group: The patients were included if they were of 18 years or older, with a diagnosis of diabetes mellitus for more than three years.
  Interventions: Diagnostic Test: Evaluation of biomechanics and viscoelastic properties of plantar fascia
- NonDiabetic Group: The healthy age-matched control group was included.
  Interventions: Diagnostic Test: Evaluation of biomechanics and viscoelastic properties of plantar fascia

INTERVENTIONS:
Diagnostic Test: Evaluation of biomechanics and viscoelastic properties of plantar fascia — The biomechanical and viscoelastic properties of the plantar fascia will be measured with the MyotonPRO device.
  Other Names: Falls Efficacy Scale

SUMMARY:
In this study, an attempt has been made to analyze the changes in soft tissue biomechanical properties of plantar surface in diabetes. The second aim of this study was to explore the relationships between fear of falling, physical performance, and plantar stiffness in patients with diabetes.

DETAILED DESCRIPTION:
Chronic diabetes can lead to ulceration in the plantar region and may result in amputation. Diabetes-related foot ulcerations are one of the most challenging complications of diabetes mellitus. Myotonometry, a technique to measure dynamic stiffness is preferred due to its noninvasiveness, easy employability, and rapid investigation. In this study, an attempt has been made to analyze the changes in soft tissue biomechanical properties of the plantar surface in diabetes. Increased plantar tissue stiffness is thought to alter the distribution of tensile stresses in the plantar soft tissues during gait. Combined with a reduction in plantar tissue thickness, these changes could collectively decrease the mechanical loads required to initiate soft tissue breakdown and thus lead to foot ulceration formation. Diabetes mellitus is a significant risk factor for falls in adults and is associated with an increase in fear of falling. Microvascular complications associated with DM result in multiple impairments including sensory deficits and muscle weakness due to peripheral neuropathy, loss of visual acuity due to retinopathy, and impaired postural control and falls due to vestibulopathy. The prevalence of falls and fear of falling are significantly higher in adults with diabetes mellitus. Assessment of mechanical properties of plantar tissues can aid in the early diagnosis of ulceration. In this study, an attempt has been made to analyze the changes in soft tissue biomechanical properties of the plantar surface in diabetes. The second aim of this study was to explore the relationships between fear of falling, physical performance, and plantar stiffness in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus for more than three years
* Individuals without a history of diabetes mellitus affirmed by a normal range of fasting blood sugar and hemoglobin A1C levels.
* Age≥18 years

Exclusion Criteria:

* History of central nervous system conditions
* No visual and vestibular impairments
* Amputation of the lower limb
* History of fracture
* Surgery of lumbar and lower limb
* Having pain resulting in movement difficulty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of diabetes mellitus for more than three years or individuals without a history of diabetes mellitus affirmed by a normal range of fasting blood sugar and hemoglobin A1C levels.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Biomechanical and Viscoelastic Properties | Day 1.
  The biomechanical and viscoelastic properties of the plantar fascia will be measured with MyotonPRO device. The MyotonPRO (Tallin, Estonia) is a portable hand-held myotonometer. This device is non-invasive and provides a quantitative assessment of a muscle's viscoelastic properties. These properties are characterized by different parameters such as tone, elasticity, and stiffness. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph.

SECONDARY OUTCOMES:
Fear of Falling | Day 1.
  Fear of falling will be assessed using the Falls Efficacy Scale International questionnaire. In this scale, scores are treated as continuous variables ranging from 16 to 64, where 16 indicates no concern and 64 indicates severe concern about falling. Participants in this study were further classified as having had low concern (score of 16-19), moderate concern (score of 20-27), or high concern (score ≥28) about falling.
Lower Limb Function | Day 1.
  The Short Physical Performance Battery will be used for Lower limb function assessment. It is an objective measure of lower-extremity function that includes 4-meter gait speed at usual pace, three standing balance tests, and time to complete five chair rises Composite scores range from 0 to 12 with higher scores reflecting better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Hospital, Istanbul, Turkey (Türkiye)